CLINICAL TRIAL: NCT05993052
Title: Neutrophil-Lymphocyte Ratio and Carotid Plaque Burden in Patients With Philadelphia Negative Myeloproliferative Neoplasms and Their Relation to JAK2V617F Mutation
Brief Title: Carotid Plaque Burden in Patients With Philadelphia Negative Myeloproliferative Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Gaber Mahmoud, Dr, Sohag University
Other Study IDs: Carotid Doppler in MPNs
Record Dates: First submitted 2023-08-06; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In around 90% of the patients with MPNs, an acquired mutation that promotes JAK/STAT signaling is identified [3, 4]. The JAK/STAT pathway transduces signals from cytokines including erythropoietin, thrombopoietin, and granulocyte colony-stimulating factor.24 A point mutation that activates JAK2, JAK2V617F, is present in around 95% of patients with PV and 40% to 60% of patients with ET and MF

DETAILED DESCRIPTION:
All patients will be subjected to a thorough assessment of history, complete clinical examination, and investigations as complete blood picture including neutrophil-lymphocyte ratio which will be analyzed with automated blood count analyzers, serum uric acid, serum creatinine and lipid profile. All patients will undergo carotid imaging using Colour Doppler ultrasonography for assessment of carotid plaque burden.

The control group will undergo carotid ultrasonography who will be recruited among apparently healthy volunteers aiming to match the patient group regarding age, sex and classical risk factors for atherosclerosis as arterial hypertension, hyperlipidemia, diabetes, smoking or obesity.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older who were newly diagnosed to have Philadelphia negative myeloproliferative neoplasms between September 2014 and November 2022 at Sohag university hospital, department of internal medicine, hematology unit and hematology outpatient clinic.

Exclusion Criteria:

* Patients were excluded if: (1) their disease of thrombocytosis or polycythemia was determined to be reactive, (2) their disease was not newly diagnosed, (3) their disease met WHO criteria for chronic or acute myeloid leukemia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with Philadelphia negative myeloproliferative neoplasms who were diagnosed according to the WHO 2016 criteria, at Sohag university hospital, department of internal medicine, hematology unit and hematology outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Neutrophil-Lymphocyte Ratio in Patients with Philadelphia Negative Myeloproliferative Neoplasms | baseline
  All patients will be subjected to a thorough assessment of history, complete clinical examination, and investigations as complete blood picture including neutrophil-lymphocyte ratio which will be analyzed with automated blood count analyzers, serum uric acid, serum creatinine and lipid profile.
Carotid Plaque Burden in Patients with Philadelphia Negative Myeloproliferative Neoplasms | baseline
  All patients will undergo carotid imaging using Colour Doppler ultrasonography for assessment of carotid plaque burden. Extracranial carotid arteries were divided into three sectors on each side: common carotid artery and its bulb, internal carotid artery, and external carotid artery. At least one plaque in any sector was scored 1 point, while the absence of plaques was scored 0. Thus, the carotid plaque score ranged from 0 (absence of plaques) to 6 (plaques in all sectors)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Gaber, Principal Investigator — Sohag University
Locations (1):
- Faculty of Medicine, Sohag, Egypt

REFERENCES:
- [Background] Accorsi F. Color Doppler of the extracranial and intracranial arteries in the acute phase of cerebral ischemia. J Ultrasound. 2013 Sep 21;16(4):187-93. doi: 10.1007/s40477-013-0036-7. eCollection 2013 Sep 21. PMID 24432173
- [Background] Kralovics R, Passamonti F, Buser AS, Teo SS, Tiedt R, Passweg JR, Tichelli A, Cazzola M, Skoda RC. A gain-of-function mutation of JAK2 in myeloproliferative disorders. N Engl J Med. 2005 Apr 28;352(17):1779-90. doi: 10.1056/NEJMoa051113. PMID 15858187